CLINICAL TRIAL: NCT03402360
Title: Effectiveness of Virtual Environment Rehabilitation in Patients With Acquired Brain Injury: Clinical Randomized Controlled Trial
Brief Title: Virtual Reality Rehabilitation in Patients With Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Sandro Iannaccone, Head of Neuro Rehabilitation Unit, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR-ABI
Record Dates: First submitted 2018-01-09; First posted 2018-01-18 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Acquired Brain Injury
Keywords: Virtual Reality; Rehabilitation; Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality rehabilitation group (Experimental): The Virtual Reality group will perform upper extremity motor rehabilitation and neurocognitive rehabilitation based on virtual reality training.
  Interventions: Other: Virtual Reality rehabilitation group
- Control group (Active Comparator): The Control group will perform the same motor and neurocognitive rehabilitation but with the virtual reality turned off.
  Interventions: Other: Control group rehabilitation

INTERVENTIONS:
Other: Virtual Reality rehabilitation group — Three hours rehabilitation sessions every day that will consist in two hours of physiotherapy and one hour of neurocognitive rehabilitation, for 15 consecutive working days (3 weeks).
  1 hour: conventional physiotherapy
  1 hour: virtual reality upper extremity motor rehabilitation
  1 hour: virtual reality neurocognitive training
  Arms: Virtual Reality rehabilitation group
Other: Control group rehabilitation — Three hours rehabilitation sessions every day that will consist in two hours of physiotherapy and one hour of neurocognitive rehabilitation, for 15 consecutive working days (3 weeks).
  1 hour: conventional physiotherapy
  1 hour: upper extremity motor rehabilitation
  1 hour: neurocognitive training
  Arms: Control group

SUMMARY:
The aim of the study is to investigate the effectiveness of motor and cognitive virtual environment rehabilitation on upper limb function in sub-acute patients after an acquired brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Acquired Brain Injury within 1 month before the recruitment;
* Score between 0 and 3 at the Motor Arm subscore of the Italian version of the National Institutes of Health Stroke Scale (it-NIHSS);
* Score between 9 and 15 at the Glasgow Coma Scale for the traumatic brain injury Acquired Brain Injury.

Exclusion Criteria:

* Denial of informed consent;
* Visual deficits that interfere with the virtual reality rehabilitation;
* Score under 18 at the Mini Mental State Examination;
* Severe orthopedic deficit;
* Patients with pace maker;
* Patients with contraindication to undergo magnetic resonance;
* Pregnant women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Upper Extremity (FMUE) | From Baseline (T0) to 3 weeks of rehabilitation (T1)
  Items are scored on a 3-point ordinal scale
  0 = cannot perform; 1 = performs partially; 2 = performs fully.
  Maximum Score = 66 points

SECONDARY OUTCOMES:
Change in Action Research Arm Test (ARAT) | From Baseline (T0) to 3 weeks of rehabilitation (T1)
Change in Functional Independence Measures (FIM) | From Baseline (T0) to 3 weeks of rehabilitation (T1)
Change in Mini Mental State Examination (MMSE) | From Baseline (T0) to 3 weeks of rehabilitation (T1)
Change in Montreal Cognitive Assessment (MoCA) | From Baseline (T0) to 3 weeks of rehabilitation (T1)
Change in Beck Depression Inventory (BDI) | From Baseline (T0) to 3 weeks of rehabilitation (T1)
Change in 36-Item Short Form Survey (SF-36) | From Baseline (T0) to 3 weeks of rehabilitation (T1)

OTHER OUTCOMES:
Change in Resting state functional MRI (fMRI) | From Baseline (T0) to 3 weeks of rehabilitation (T1)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCSS Ospedale San Raffaele, Milan, MI, Italy